CLINICAL TRIAL: NCT03256955
Title: The Comparison of the TOF Cuff Monitor® With the TOF Watch SX® Monitor:
Brief Title: Validation of the TOF Cuff Monitor® Which Measures Neuromuscular Block on the Upper Arm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christoph Czarnetzki (Other)
Responsible Party: Sponsor-Investigator, Christoph Czarnetzki, Médecin adjoint, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TofCuff Study
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Neuromuscular Blockade
Keywords: Validation study for a neuromuscular monitoring device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tof Watch SX and Tof Cuff (Other): Patients undergoing surgery with intubation and receiving a single intubation dose of rocuronium (0.6 mg/kg) under propofol anesthesia will have monitoring of neuromuscular block with two monitors simultaneously.
  Interventions: Device: Tof cuff; Device: Tof Watch SX

INTERVENTIONS:
Device: Tof cuff — The Tof Cuff will be installed on one arm. After anesthesia induction the Tof Cuff will be calibrated and continuos monitoring of the neuromuscular block started until complete recovery of neuromuscular block.
Device: Tof Watch SX — The Tof Watch SX will be installed on the opposite arm to the Tof Cuff. After anesthesia induction the Tof Watch SX will be calibrated and continuos monitoring of the neuromuscular block started until complete recovery of neuromuscular block.

SUMMARY:
Neuromuscular blocking agents (NMBAs) are frequently used in anesthesia and quantitative neuromuscular monitoring is standard care. The TOF WATCH SX® monitor is considered as one of the reference monitoring devices in clinical research and clinical practice. With this monitor the ulnar nerve is stimulated at the wrist and the force of the movement of the thumb is measured with acceleromyography. This method requires freedom of movement of the patient's thumb. Unfortunately this is not always possible due to the constraints of patient positioning during the operation. The TOF Cuff® monitor is a modified non-invasive blood pressure cuff that incorporates stimulating electrodes in its inner surface and is based on the stimulation of the peripheral nerve in the arm (brachial plexus, ulnar and median nerves principally). The evoked neuromuscular activity is recorded through the changes in pressure generated in the inner part of the cuff by the muscular activity after the stimulus. Moreover, this device can be used for non-invasive reading of the blood pressure. This device has been validated with mechanomyography, but was never been compared with acceleromyography, which is the most common used neuromuscular monitoring method.

DETAILED DESCRIPTION:
Neuromuscular blocking agents (NMBAs) are frequently used in anesthesia for tracheal intubation, artificial ventilation, and continued muscle relaxation during surgical interventions. It is of particular importance to measure the neuromuscular block for several reasons:

1. To monitor the onset of neuromuscular block and to intubate when deep muscular relaxation is attained.
2. To choose the best antagonist and its dosage dependent of the degree of neuromuscular block (for instance sugammadex for deep neuromuscular block or neostigmine for superficial block).
3. To avoid antagonization of neuromuscular block in the case of complete recovery of neuromuscular function.

It is proven that monitoring of neuromuscular block reduces patient mortality. It avoids postoperative residual curarization, which is associated with complications such as hypoxemia, bronchoaspiration and pneumonia. Therefore the development and validation of new and efficacious neuromuscular monitoring devices is of great importance.

Neuromuscular monitoring is done by stimulating with an electric current a nerve and to measure the response of the corresponding muscle. In clinical practice acceleromyography is the most often used quantitative measurement method, because it is much easier to apply than other established quantitative neuromuscular monitoring methods such as mechanomyograpy and electromyography. Acceleromyography is based on the piezoelectric effect where mechanical forces at play on the surfaces of certain materials, such as crystals or ceramics, induce an electrical current. According to Newton's second law of motion, force equals mass times acceleration (F=m x a). At constant mass, the acceleration measured and the voltage thereby generated can be used to derive the force of the stimulated muscle. It is standard practice to stimulate the ulnar nerve at the wrist and to measure the movement of the adductor pollicis. In the research setting acceleromyography (TOF Watch SX® monitor) is an established and widely used method. This method requires freedom of movement of the patient's thumb. Unfortunately this is not always possible due to the constraints of patient positioning during the operation. The TOF Cuff® monitor is a modified non-invasive blood pressure cuff that incorporates stimulating electrodes in its inner surface and is based on the stimulation of the peripheral nerve in the arm (brachial plexus, ulnar and median nerves principally). The evoked neuromuscular activity is recorded through the changes in pressure generated in the inner part of the cuff by the muscular activity after the stimulus. Moreover, this device can be used for non-invasive reading of the blood pressure. This device has been validated with mechanomyography, but was never been compared with acceleromyography, which is the most common used neuromuscular monitoring method.

ELIGIBILITY:
Inclusion Criteria:

* Patients, age ≥18 to 65 years
* Patient with American Society of Anesthesiology [ASA] status I or II
* Patient able to read and understand the information sheet and to sign and date the consent form
* Patient scheduled for elective surgery lasting at least 60 minutes

Exclusion Criteria:

* Patient with a history of allergy or hypersensitivity to rocuronium
* Patient with pacemaker
* Patients with neuromuscular disease
* Patients with preoperative medications known to influence neuromuscular function (for instance aminoglycosides, phenytoin, lidocaine)
* Patients with electrolyte abnormalities (for instance, hypermagnesemia)
* Patients with a body mass index <19 or >30 kg m2
* Patient having participated in any clinical trial within 30 days, inclusive, of signing the informed consent form of the current trial
* Patients undergoing interventions that need a continuous deep NMB (for surgical reasons).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Total recovery time of neuromuscular block | 60 to 120 minutes
  The total recovery time, i.e. total duration of the neuromuscular block is defined as the time in minutes from start of injection of rocuronium until a normalized TOF ratio of 90% (Dur TOF 0.9). TOF = Train of Four

SECONDARY OUTCOMES:
Onset time | 1 to 4 minutes
  time in seconds from start of injection of rocuronium until 95% depression of the first twitch (T1) of the TOF(Train of Four)
Duration TOF count 1 | 20 - 30 minutes
  Time (in minutes) from administration of rocuronium to emergence of the 1st twitch of the TOF (Dur TOFc1)
Duration TOF 25% | 30 - 40 minutes
  Time (in minutes) from administration of rocuronium to emergence of a normalized TOF ratio of 25%
Duration TOF 50% | 30 - 50 minutes
  Time (in minutes) from administration of rocuronium to emergence of a normalized TOF ratio of 50%
Duration TOF 75% | 30 - 60 minutes
  Time (in minutes) from administration of rocuronium to emergence of a normalized TOF ratio of 75%

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Czarnetzki, MD, Study Chair — University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

REFERENCES:
- [Background] Rodiera J, Serradell A, Alvarez-Gomez JA, Aliaga L. The cuff method: a pilot study of a new method of monitoring neuromuscular function. Acta Anaesthesiol Scand. 2005 Nov;49(10):1552-8. doi: 10.1111/j.1399-6576.2005.00777.x. PMID 16223405
- [Background] Veiga Ruiz G, Garcia Cayuela J, Orozco Montes J, Parreno Caparros M, Garcia Rojo B, Aguayo Albasini JL. Monitoring intraoperative neuromuscular blockade and blood pressure with one device (TOF-Cuff): A comparative study with mechanomyography and invasive blood pressure. Rev Esp Anestesiol Reanim. 2017 Dec;64(10):560-567. doi: 10.1016/j.redar.2017.03.013. Epub 2017 Jun 27. English, Spanish. PMID 28662770
- [Result] Sfeir Machado E, Keli-Barcelos G, Dupuis-Lozeron E, Tramer MR, Czarnetzki C. Assessment of spontaneous neuromuscular recovery: A comparison of the TOF-Cuff(R) with the TOF Watch SX(R). Acta Anaesthesiol Scand. 2020 Feb;64(2):173-179. doi: 10.1111/aas.13487. Epub 2019 Oct 28. PMID 31593293
- See also: Thesis for the validation of the tof cuff (in spanish) — http://www.tdx.cat/handle/10803/307220